CLINICAL TRIAL: NCT05972265
Title: Exercise and Cognition in Middle-Aged Adults With Histories of Childhood Trauma and Cognitive Complaints
Brief Title: Childhood Trauma, Exercise, and Cognition
Acronym: CTEC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Erin Logue, assistant professor, University of Texas at Austin
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: STUDY00004558
Record Dates: First submitted 2023-07-03; First posted 2023-08-02 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Adverse Childhood Experiences
MeSH Terms: interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Acute Exercise Moderate first (Experimental): Day 1 Assessments, Day 8 Moderate Intensity Exercise (followed by symptom measures and neuropsychological tests), Day 15 Light Intensity Exercise (symptom measures and neuropsychological tests)
  Interventions: Behavioral: Moderate Intensity Exercise (one day); Behavioral: Placebo - Light Intensity Exercise (one day); Other: Day 1 Assessments; Other: Symptom Measures and Neuropsychological Tests
- Acute Exercise Light first (Active Comparator): Control Day 1 Assessments (symptom measures, neuropsychological tests, and cognitive complaints interview), Day 8 Light Intensity Exercise (followed by symptom measures and neuropsychological tests), Day 15 Moderate Intensity Exercise (symptom measures and neuropsychological tests)
  Interventions: Behavioral: Moderate Intensity Exercise (one day); Behavioral: Placebo - Light Intensity Exercise (one day); Other: Day 1 Assessments; Other: Symptom Measures and Neuropsychological Tests
- Chronic Exercise Moderate (Experimental): 9-weeks Moderate Intensity Exercise Day 36 (at 3 weeks) Assessments Day 57 (at 6 weeks) Assessments Day 78 (at 9 weeks) Assessments
  Interventions: Behavioral: Moderate Intensity Exercise (9 wks); Other: Day 36 Assessments; Other: Day 57 Assessments; Other: Day 78 Assessments
- Activity as Usual (No Intervention): 9-week activity as usual Day 36 (at 3 weeks) Assessments Day 57 (at 6 weeks) Assessments Day 78 (at 9 weeks) Assessments

INTERVENTIONS:
Behavioral: Moderate Intensity Exercise (one day) — Participants will engage in 40 minutes of cycling at 70-75% maximum heart rate (MHR).
  Arms: Acute Exercise Light first; Acute Exercise Moderate first
Behavioral: Placebo - Light Intensity Exercise (one day) — Control participants will engage in 40 minutes cycling at 40-50% maximum heart rate (MHR).
  Arms: Acute Exercise Light first; Acute Exercise Moderate first
Behavioral: Moderate Intensity Exercise (9 wks) — Participants will be asked to engage in moderate-intensity activity four days each week, 40 minutes each time, and will wear an activity monitoring device to assess their fidelity to the intervention.
  Arms: Chronic Exercise Moderate
Other: Day 1 Assessments — Cognitive complaints interview, Center for Epidemiological Studies Depression Scale Revised (CESD-R), Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5), Life Events Checklist (LEC-5), and neuropsychological testing: approximately 1.50 hours
  Arms: Acute Exercise Light first; Acute Exercise Moderate first
Other: Symptom Measures and Neuropsychological Tests — Center for Epidemiological Studies Depression Scale Revised (CESD-R), Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5), and neuropsychological testing: approximately 1.25 hours
  Arms: Acute Exercise Light first; Acute Exercise Moderate first
Other: Day 36 Assessments — Activity monitoring device charged and data downloaded, questions regarding fidelity to activity as usual or moderate-intensity exercise and any difficulties, Cognitive complaints interview, Center for Epidemiological Studies Depression Scale Revised (CESD-R), Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5), neuropsychological testing, and activity monitoring device returned to participant: approximately 2.00 hours
  Arms: Chronic Exercise Moderate
Other: Day 57 Assessments — Activity monitoring device charged and data downloaded, questions regarding fidelity to activity as usual or moderate-intensity exercise and any difficulties, Cognitive complaints interview, Center for Epidemiological Studies Depression Scale Revised (CESD-R), Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5), neuropsychological testing, and activity monitoring device returned to participant: approximately 2.00 hours
  Arms: Chronic Exercise Moderate
Other: Day 78 Assessments — Activity monitoring device charged and data downloaded, questions regarding fidelity to activity as usual or moderate-intensity exercise and any difficulties, Cognitive complaints interview, Center for Epidemiological Studies Depression Scale Revised (CESD-R), Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5), neuropsychological testing, and activity monitoring device returned to participant: approximately 2.00 hours
  Arms: Chronic Exercise Moderate

SUMMARY:
This study aims to identify and compare the effects of acute and chronic exercise interventions on cognition in middle-aged adults with cognitive complaints and a history of abuse or neglect in childhood. Each participant will be enrolled in the study for up to 78 days, in five parts following verification that the participant meets criteria to be included in the study: 1) initial assessment; 2) first acute exercise condition in lab, symptom measures, and neuropsychological testing; 3) second acute exercise condition in lab, symptom measures, and neuropsychological testing; and 4) 9-week exercise intervention or activity as usual outside of lab, with interview, symptom measures, and neuropsychological testing at three-week intervals.

ELIGIBILITY:
Inclusion Criteria:

* between 40 and 60 years of age
* history of child abuse or neglect
* have a complaint about memory, attention, or executive function
* native or fluent English speaker
* normal or corrected to normal vision and hearing
* medically healthy

Exclusion Criteria:

* Score indicating a history of moderate-intensity activity, hard-intensity activity, or very-hard intensity activity on the Stanford Brief Activity Survey
* current excessive alcohol or other substance use
* eating disorder, bipolar disorder, schizophrenia spectrum disorders, or those judged to be an immediate suicide risk based on having an active plan with intent
* autism spectrum disorder, attention-deficit/hyperactivity disorder (ADHD), or other neurodevelopmental disorder
* neurocognitive disorder, or illnesses or history of neurological events known to cause neurocognitive disorders (e.g., traumatic brain injury, status epilepticus, stroke)
* reported chest pain or dizziness during exercise; any endorsed and not controlled medical condition that could make exercise contraindicated, including hypertension; heart disease; heart failure; hear rhythm disorders; heart valve disease; metabolic conditions; chronic obstructive pulmonary disease; pulmonary hypertension; cystic fibrosis; asthma; and bone, joint, or soft tissue problems
* pregnancy, major medical disorders such as cancer, or any other condition believed to put a participant at risk

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-12-04 (Estimated); Study Completion 2024-12-04 (Estimated)

PRIMARY OUTCOMES:
Change in performance (i.e., raw score of number of words recalled, in whole numbers) on the Loewenstein-Acevedo Scales for Semantic Interference and Learning (LASSI-L) from baseline will be compared within subjects. | one week before first acute exercise condition (baseline), after acute exercise condition on day 8, and after acute exercise condition on day 15.
  The Loewenstein-Acevedo Scales for Semantic Interference and Learning (LASSI-L) is a reliable, well-validated measure of verbal learning and memory. The minimum score on this measure is 0, and the highest score is 15. Higher scores indicate better memory.
Change in performance (i.e., raw score of total correct, in whole numbers) on the Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV) Digit Span test from baseline will be compared within subjects. | one week before first acute exercise condition (baseline), after acute exercise condition on day 8, and after acute exercise condition on day 15
  The Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV) Digit Span test is a reliable, well-validated measure of auditory attention and working memory. The minimum score on this measure is 0, and the highest score is 48. Higher scores indicate better attention.
Change in performance (i.e., raw scores of time to complete task, in seconds) on the Trail Making Test (TMT) from baseline will be compared within subjects. | exercise condition on day 8, and after acute exercise condition on day 15
  The Trail Making Test (TMT) is a reliable, well-validated measure of visual attention, processing speed, and executive function. The minimum score on this measure is 1, and the highest score is 300. Lower scores indicate better executive function.
Change in performance (i.e., raw scores of time to complete task, in seconds) on the Symbol Digit Modalities Test (SDMT) from baseline will be compared within subjects. | one week before first acute exercise condition (baseline), after acute exercise condition on day 8, and after acute exercise condition on day 15
  The Symbol Digit Modalities Test (SDMT) is a reliable, well-validated measure of visual working memory, processing speed, and executive function. The minimum score on this measure is 0, and the highest score is 110. Higher scores indicate faster processing speed.
Change in performance (i.e., raw score of total correct, in whole numbers) on the Paced Auditory Serial Addition Test (PASAT) from baseline will be compared within subjects. | one week before first acute exercise condition (baseline), after acute exercise condition on day 8, and after acute exercise condition on day 15
  The Paced Auditory Serial Addition Test (PASAT) is a reliable, well-validated measure of auditory working memory, processing speed, and executive function. The minimum score on this measure is 0, and the highest score is 60. Higher scores indicate better working memory.
Change in performance (i.e., raw scores of total words generated, in whole numbers) on the Controlled Oral Word Association Test (COWAT) from baseline will be compared within subjects. | one week before first acute exercise condition (baseline), after acute exercise condition on day 8, and after acute exercise condition on day 15
  The Controlled Oral Word Association Test (COWAT) is a reliable, well-validated measure of language and executive function. The minimum score on this measure is 0, and the highest score is 180. Higher scores indicate better ability to generate words given a phonemic cue.
Change from baseline performance (i.e., raw score of number of words recalled, in whole numbers) on the Loewenstein-Acevedo Scales for Semantic Interference and Learning (LASSI-L) at 3 weeks post-chronic exercise intervention. | one week before first acute exercise condition (baseline) and after 3 weeks of the chronic exercise condition or activity as usual
  Assessed between participants assigned to 9-week intervention and those assigned to activity as usual. The Loewenstein-Acevedo Scales for Semantic Interference and Learning (LASSI-L) is a reliable, well-validated measure of verbal learning and memory. The minimum score on this measure is 0, and the highest score is 15. Higher scores indicate better memory.
Change from baseline performance (i.e., raw score of total correct, in whole numbers) on the Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV) Digit Span test at 3 weeks post-chronic exercise intervention. | one week before first acute exercise condition (baseline) and after 3 weeks of the chronic exercise condition or activity as usual
  Assessed between participants assigned to 9-week intervention and those assigned to activity as usual. The Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV) Digit Span test is a reliable, well-validated measure of auditory attention and working memory. The minimum score on this measure is 0, and the highest score is 48. Higher scores indicate better attention.
Change from baseline performance (i.e., raw scores of time to complete task, in seconds) on the Trail Making Test (TMT) at 3 weeks post-chronic exercise intervention. | one week before first acute exercise condition (baseline) and after 3 weeks of the chronic exercise condition or activity as usual
  Assessed between participants assigned to 9-week intervention and those assigned to activity as usual. The Trail Making Test (TMT) is a reliable, well-validated measure of visual attention, processing speed, and executive function. The minimum score on this measure is 1, and the highest score is 300. Lower scores indicate better executive function.
Change from baseline performance (i.e., raw scores of time to complete task, in seconds) on the Symbol Digit Modalities Test (SDMT) at 3 weeks post-chronic exercise intervention. | one week before first acute exercise condition (baseline) and after 3 weeks of the chronic exercise condition or activity as usual
  Assessed between participants assigned to 9-week intervention and those assigned to activity as usual. The Symbol Digit Modalities Test (SDMT) is a reliable, well-validated measure of visual working memory, processing speed, and executive function. The minimum score on this measure is 0, and the highest score is 110. Higher scores indicate faster processing speed.
Change from baseline performance (i.e., raw score of total correct, in whole numbers) on the Paced Auditory Serial Addition Test (PASAT) at 3 weeks post-chronic exercise intervention. | one week before first acute exercise condition (baseline) and after 3 weeks of the chronic exercise condition or activity as usual
  Assessed between participants assigned to 9-week intervention and those assigned to activity as usual. The Paced Auditory Serial Addition Test (PASAT) is a reliable, well-validated measure of auditory working memory, processing speed, and executive function. The minimum score on this measure is 0, and the highest score is 60. Higher scores indicate better working memory.
Change from baseline performance (i.e., raw scores of total words generated, in whole numbers) on the Controlled Oral Word Association Tet (COWAT) at 3 weeks post-chronic exercise intervention. | one week before first acute exercise condition (baseline) and after 3 weeks of the chronic exercise condition or activity as usual
  Assessed between participants assigned to 9-week intervention and those assigned to activity as usual. The Controlled Oral Word Association Test (COWAT) is a reliable, well-validated measure of language and executive function. The minimum score on this measure is 0, and the highest score is 180. Higher scores indicate better ability to generate words given a phonemic cue.
Change from baseline performance (i.e., raw score of number of words recalled, in whole numbers) on the Loewenstein-Acevedo Scales for Semantic Interference and Learning (LASSI-L) at 6 weeks post-chronic exercise intervention. | one week before first acute exercise condition (baseline) and after 6 weeks of the chronic exercise condition or activity as usual
  Assessed between participants assigned to 9-week intervention and those assigned to activity as usual. The Loewenstein-Acevedo Scales for Semantic Interference and Learning (LASSI-L) is a reliable, well-validated measure of verbal learning and memory. The minimum score on this measure is 0, and the highest score is 15. Higher scores indicate better memory.
Change from baseline performance (i.e., raw score of total correct, in whole numbers) on the Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV) Digit Span test at 6 weeks post-chronic exercise intervention. | one week before first acute exercise condition (baseline) and after 6 weeks of the chronic exercise condition or activity as usual
  Assessed between participants assigned to 9-week intervention and those assigned to activity as usual. The Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV) Digit Span test is a reliable, well-validated measure of auditory attention and working memory. The minimum score on this measure is 0, and the highest score is 48. Higher scores indicate better attention.
Change from baseline performance (i.e., raw scores of time to complete task, in seconds) on the Trail Making Test (TMT) at 6 weeks post-chronic exercise intervention. | one week before first acute exercise condition (baseline) and after 6 weeks of the chronic exercise condition or activity as usual
  Assessed between participants assigned to 9-week intervention and those assigned to activity as usual. The Trail Making Test (TMT) is a reliable, well-validated measure of visual attention, processing speed, and executive function. The minimum score on this measure is 1, and the highest score is 300. Lower scores indicate better executive function.
Change from baseline performance (i.e., raw scores of time to complete task, in seconds) on the Symbol Digit Modalities Test (SDMT) at 6 weeks post-chronic exercise intervention. | one week before first acute exercise condition (baseline) and after 6 weeks of the chronic exercise condition or activity as usual
  Assessed between participants assigned to 9-week intervention and those assigned to activity as usual. The Symbol Digit Modalities Test (SDMT) is a reliable, well-validated measure of visual working memory, processing speed, and executive function. The minimum score on this measure is 0, and the highest score is 110. Higher scores indicate faster processing speed.
Change from baseline performance (i.e., raw score of total correct, in whole numbers) on the Paced Auditory Serial Addition Test (PASAT) at 6 weeks post-chronic exercise intervention. | one week before first acute exercise condition (baseline) and after 6 weeks of the chronic exercise condition or activity as usual
  Assessed between participants assigned to 9-week intervention and those assigned to activity as usual. The Paced Auditory Serial Addition Test (PASAT) is a reliable, well-validated measure of auditory working memory, processing speed, and executive function. The minimum score on this measure is 0, and the highest score is 60. Higher scores indicate better working memory.
Change from baseline performance (i.e., raw scores of total words generated, in whole numbers) on the Controlled Oral Word Association Tet (COWAT) at 6 weeks post-chronic exercise intervention. | one week before first acute exercise condition (baseline) and after 6 weeks of the chronic exercise condition or activity as usual
  Assessed between participants assigned to 9-week intervention and those assigned to activity as usual. The Controlled Oral Word Association Test (COWAT) is a reliable, well-validated measure of language and executive function. The minimum score on this measure is 0, and the highest score is 180. Higher scores indicate better ability to generate words given a phonemic cue.
Change from baseline performance (i.e., raw score of number of words recalled, in whole numbers) on the Loewenstein-Acevedo Scales for Semantic Interference and Learning (LASSI-L) at 9 weeks post-chronic exercise intervention. | one week before first acute exercise condition (baseline) and after 9 weeks of the chronic exercise condition or activity as usual
  Assessed between participants assigned to 9-week intervention and those assigned to activity as usual. The Loewenstein-Acevedo Scales for Semantic Interference and Learning (LASSI-L) is a reliable, well-validated measure of verbal learning and memory. The minimum score on this measure is 0, and the highest score is 15. Higher scores indicate better memory.
Change from baseline performance (i.e., raw score of total correct, in whole numbers) on the Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV) Digit Span test at 9 weeks post-chronic exercise intervention. | one week before first acute exercise condition (baseline) and after 9 weeks of the chronic exercise condition or activity as usual
  Assessed between participants assigned to 9-week intervention and those assigned to activity as usual. The Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV) Digit Span test is a reliable, well-validated measure of auditory attention and working memory. The minimum score on this measure is 0, and the highest score is 48. Higher scores indicate better attention.
Change from baseline performance (i.e., raw scores of time to complete task, in seconds) on the Trail Making Test (TMT) at 9 weeks post-chronic exercise intervention. | one week before first acute exercise condition (baseline) and after 9 weeks of the chronic exercise condition or activity as usual
  Assessed between participants assigned to 9-week intervention and those assigned to activity as usual. The Trail Making Test (TMT) is a reliable, well-validated measure of visual attention, processing speed, and executive function. The minimum score on this measure is 1, and the highest score is 300. Lower scores indicate better executive function.
Change from baseline performance (i.e., raw scores of time to complete task, in seconds) on the Symbol Digit Modalities Test (SDMT) at 9 weeks post-chronic exercise intervention. | one week before first acute exercise condition (baseline) and after 9 weeks of the chronic exercise condition or activity as usual
  Assessed between participants assigned to 9-week intervention and those assigned to activity as usual. The Symbol Digit Modalities Test (SDMT) is a reliable, well-validated measure of visual working memory, processing speed, and executive function. The minimum score on this measure is 0, and the highest score is 110. Higher scores indicate faster processing speed.
Change from baseline performance (i.e., raw score of total correct, in whole numbers) on the Paced Auditory Serial Addition Test (PASAT) at 9 weeks post-chronic exercise intervention. | one week before first acute exercise condition (baseline) and after 9 weeks of the chronic exercise condition or activity as usual
  Assessed between participants assigned to 9-week intervention and those assigned to activity as usual. The Paced Auditory Serial Addition Test (PASAT) is a reliable, well-validated measure of auditory working memory, processing speed, and executive function. The minimum score on this measure is 0, and the highest score is 60. Higher scores indicate better working memory.
Change from baseline performance (i.e., raw scores of total words generated, in whole numbers) on the Controlled Oral Word Association Tet (COWAT) at 9 weeks post-chronic exercise intervention. | one week before first acute exercise condition (baseline) and after 9 weeks of the chronic exercise condition or activity as usual
  Assessed between participants assigned to 9-week intervention and those assigned to activity as usual. The Controlled Oral Word Association Test (COWAT) is a reliable, well-validated measure of language and executive function. The minimum score on this measure is 0, and the highest score is 180. Higher scores indicate better ability to generate words given a phonemic cue.
Change from baseline cognitive complaints (i.e., total number of complaints) at 3 weeks post-chronic exercise intervention. | one week before first acute exercise condition (baseline) and after 3 weeks of the chronic exercise condition or activity as usual
  Assessed between participants assigned to 9-week intervention and those assigned to activity as usual. To assess cognitive complaints, an interview by the primary investigator, asking about symptoms of difficulties with attention, thinking speed, language, memory, and executive function.
Change from baseline cognitive complaints (i.e., total number of complaints) at 6 weeks post-chronic exercise intervention. | one week before first acute exercise condition (baseline) and after 6 weeks of the chronic exercise condition or activity as usual
  Assessed between participants assigned to 9-week intervention and those assigned to activity as usual. To assess cognitive complaints, an interview by the primary investigator, asking about symptoms of difficulties with attention, thinking speed, language, memory, and executive function.
Change from baseline cognitive complaints (i.e., total number of complaints) at 9 weeks post-chronic exercise intervention. | one week before first acute exercise condition (baseline) and after 9 weeks of the chronic exercise condition or activity as usual
  Assessed between participants assigned to 9-week intervention and those assigned to activity as usual. To assess cognitive complaints, an interview by the primary investigator, asking about symptoms of difficulties with attention, thinking speed, language, memory, and executive function.

SECONDARY OUTCOMES:
Change in total score on the Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5). | one week before first acute exercise condition (baseline); after acute exercise condition on day 8; after acute exercise condition on day 15; and after 3 weeks, 6 weeks, and 9 weeks of the chronic exercise condition or activity as usual
  The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) a 20-item widely used questionnaire to assess the severity of symptoms of posttraumatic stress disorder (PTSD). The minimum score on this measure is 0, and the highest score is 80. Higher scores indicate worse symptoms of PTSD.
Change in total score on the Center for Epidemiological Studies Depression Scale Revised (CESD-R). | one week before first acute exercise condition (baseline); after acute exercise condition on day 8; after acute exercise condition on day 15; and after 3 weeks, 6 weeks, and 9 weeks of the chronic exercise condition or activity as usual
  The Center for Epidemiological Studies Depression Scale Revised (CESD-R) is a 20-item self-report measure of depression symptoms used in research. The minimum score on this measure is 0, and the highest score is 60. Higher scores indicate worse symptoms of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Logue, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No